CLINICAL TRIAL: NCT05740215
Title: A Multicenter, Open-label, Phase Ib/II Study on the Efficacy and Safety of F520 Combined With Lenvatinib in the Treatment of Patients With Advanced Solid Tumors
Brief Title: Efficacy and Safety Study of F520 Combined With Lenvatinib in the Treatment of Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-102
Record Dates: First submitted 2023-02-03; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumors
Keywords: F520; PD-1
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F520 combined with lenvatinib (Experimental): F520:
  F520 (200 mg) administered intravenously (IV) on Day 1 of each 21-day cycle in the phase Ib and II studies until progressive disease, unacceptable toxicity or ending treatment for other reasons. [Time Frame: up to 2 years post infusion]
  Lenvatinib:
  In the phase Ib study, three dose groups of 20 mg, 16 mg and 12 mg lenvatinib were designed. 3 to 6 subjects are expected to be enrolled in each dose group according to observed DLT. The designated dose of lenvatinib administered orally once daily (QD) according to the assigned dose group.
  In the phase II study, lenvatinib administered orally once daily (QD) according to recommended phase II dose (RP2D) obtained in phase Ib study.
  Interventions: Drug: F520; Drug: Lenvatinib

INTERVENTIONS:
Drug: F520 — F520 is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2)
Drug: Lenvatinib — Lenvatinib capsules

SUMMARY:
This is a multicenter, open-label, phase Ib/II study on the efficacy and safety of F520 combined with lenvatinib in the treatment of patients with advanced solid tumors. About 138~158 patients with advanced solid tumors plan to be enrolled in about 30 study sites of the study.

Part I: Phase Ib study evaluating the safety and tolerability of F520 combined with lenvatinib in patients with advanced solid tumors.

Part II: Phase II study of F520 combined with lenvatinib in endometrial cancer and cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

Phase Ib:

1. Male or female aged ≥18 years and ≤75 years old;
2. Study population: confirmed by histological and/or cytological examination patients with solid tumors (endometrial cancer, cervical cancer, non-small cell lung cancer, urothelial carcinoma, etc.), patients with metastatic solid tumors who have failed (disease progression or intolerance) after adequate standard treatment or lack effective treatments;
3. Expected survival period ≥ 12 weeks;
4. ECOG 0-1 points;
5. Blood pressure (BP) is adequately controlled with or without antihypertensive drugs, defined as BP ≤ 150/90 mmHg and unchanged antihypertensive drugs within 1 week prior to enrollment;
6. Vital organ functions meet the following requirements (Reception of granulocyte colony-stimulating factor (G-CSF) or pegylated granulocyte colony-stimulating factor (PEG-G-CSF) or blood transfusion within 14 days prior to laboratory tests is not permitted for prophylactic use):

   Blood routine: absolute neutrophil count (ANC) ≥ 1.5×109/L, hemoglobin (HGB) ≥ 90 g/L, platelet count (PLT) ≥ 75 ×109/L, lymphocyte percentage≥10%; liver function: total bilirubin level (TBIL)≤1.5×ULN, ALT and AST≤2.5×ULN; if there is liver metastasis, ALT and AST≤5×ULN; Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥40mL/min (Cr>1.5×ULN); Coagulation function: international normalized ratio (INR) ≤1.5×ULN;
7. Aagree to provide archived tumor tissue samples Or fresh tissue samples;
8. Those who understand and voluntarily sign the written informed consent.

Phase II:

1. Women aged ≥18 years and ≤75 years old;
2. Study population:

   Cohort 1: Patients with recurrent or metastatic endometrial cancer (except carcinosarcoma) who have progressed after receiving at least one line of treatment, and the number of previous platinum-containing treatment lines is ≤ 2; Cohort 2: patients with recurrent or metastatic cervical cancer (Squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma) who have progressed after receiving at least one line of platinum-containing regimens and adenosquamous carcinoma); those who progressed during or within 6 months after receiving platinum-containing regimen neoadjuvant or adjuvant chemotherapy can also be included;
3. Expected survival ≥ 12 weeks;
4. According to the RECIST1.1 standard, the subject patients must have at least one measurable target lesion (extranodal lesions: long diameter ≥ 10mm; intranodal lesions: short diameter ≥ 15mm) by enhanced CT and/or enhanced MRI;
5. ECOG 0-1 points;
6. Adequate control of blood pressure (BP) with or without antihypertensive drugs, defined as BP ≤ 150/90 mmHg and antihypertensive drugs remained unchanged within 1 week before enrollment;
7. Vital organ functions meet the following requirements (Reception of granulocyte colony-stimulating factor (G-CSF) or pegylated granulocyte colony-stimulating factor (PEG-G-CSF) or blood transfusion within 14 days prior to laboratory tests is not permitted for prophylactic use):

   Blood routine: absolute neutrophil count (ANC) ≥ 1.5×109/L, hemoglobin (HGB) ≥ 90 g/L, platelet count (PLT) ≥ 75 ×109/L, lymphocyte percentage≥10%; liver function: total bilirubin level (TBIL)≤1.5×ULN, ALT and AST≤2.5×ULN; if there is liver metastasis, ALT and AST≤5×ULN; Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥40mL/min (Cr>1.5×ULN); Coagulation function: international normalized ratio (INR) ≤1.5×ULN;
8. Those who agree to provide archived tumor tissue samples or fresh tissue samples;
9. Those who understand and voluntarily sign the written informed consent.

Exclusion Criteria:

1. Those who have received systemic tumor therapy of radiotherapy, chemotherapy, traditional Chinese medicine, hormone therapy, surgery, targeted therapy or antibody drugs within 28 days (or 5 half-lives of the drug, whichever is shorter) before the first dose; Those whose toxicity of previous anti-tumor therapy has not recovered to ≤ grade 1 (except alopecia);
2. Those who have previously received any angiogenic drugs that directly target VEGF (Subjects who have only used bevacizumab in the past can be enrolled), anti-PD-1, anti-PD-L1, anti-PD-L2 or any other Antibody or drug therapy that specifically targets T cell co-stimulation or checkpoint pathways;
3. Subjects with central nervous system (CNS) metastases, unless they have completed local therapy (eg, whole brain radiation therapy [WBRT], surgery, or radiosurgery) and have stopped corticosteroid therapy at least 4 weeks prior to the start of study treatment;
4. Inability to swallow or disease/surgery significantly affects gastrointestinal function, such as malabsorption syndrome, gastrectomy or small bowel resection, bariatric surgery, symptomatic inflammatory bowel disease, etc.;
5. Partial or complete intestinal obstruction or intestinal obstruction occurred within 1 month before the first administration;
6. Have suffered from interstitial lung disease, non-infectious pneumonia or uncontrolled lung disease in the past 3 years, including but not limited to pulmonary fibrosis, acute lung disease, etc.;
7. Those with uncontrollable or severe cardiovascular diseases, such as New York Heart Association (NYHA) congestive heart failure above grade II, unstable angina, myocardial infarction and other cardiovascular diseases occurring within 6 months before the first administration;
8. QTcF ≥ 480 milliseconds (QT interval must use Fridericia formula for heart rate correction [QTcF]);
9. Within 3 months before the first dose, there were clinically significant hematuria, hematemesis or hemoptysis (>2.5 mL red blood), or other medical history of significant bleeding (such as pulmonary hemorrhage);
10. Those with thrombosis who need treatment in the acute phase;
11. Active hepatitis patients (HBV DNA>2000 IU/mL or 1000 copies of chronic hepatitis B or chronic HBV carriers; HCV positive and HCV-RNA positive hepatitis C patients); human immunodeficiency virus (HIV) antibody positive; Treponema pallidum (TP) antibody positive;
12. Subjects with urine protein>1+ receive 24-hour urine protein quantification, urine protein ≥1g/24 hours;
13. Those with a known history of contraindications or hypersensitivity to any test drug or any known excipients;
14. Those who have had organ transplantation in the past or received autologous stem cell transplantation within 3 months before the first administration;
15. Those with a history of other malignant tumors within the past 3 years, except locally curable cancers (radical melanoma, basal or squamous cell carcinoma, carcinoma in situ of the bladder or cervix);
16. Immunosuppressant, systemic or local hormone therapy has been used within 14 days before the first administration to achieve the purpose of immunosuppression (daily dose equivalent to prednisone > 10 mg of systemic corticosteroids);
17. Those with a history of drug abuse and alcoholism within 6 months before the first administration;
18. Active autoimmune disease requiring systemic treatment within the past 2 years (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressive drugs), alternative therapy (such as physiological corticosteroid replacement therapy for thyroxine, insulin, or adrenal or pituitary insufficiency, etc.) is not considered a systemic treatment;
19. Those who received (attenuated) live vaccines within 30 days before the first administration (except for inactivated influenza vaccines such as injectable seasonal influenza vaccines and COVID-19 vaccines);
20. Pregnant or breastfeeding women, female subjects of childbearing age or male subjects whose partner is a woman of childbearing age do not agree to use highly effective methods of contraception during the study period and within 6 months after the last study drug treatment;
21. Those judged by the researchers to be unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | 21 days after first dose
  Phase Ib: The incidence of adverse events/serious adverse events, their correlation with the trial drug and their severity.
Adverse events | 21 days after first dose
  Phase Ib: The incidence of adverse events/serious adverse events, their correlation with the trial drug and their severity.
Dose-limiting toxicity (DLT) | 21 days after first dose
  Phase Ib: Assess the incidence of dose-limiting toxicity (DLT), and determine the maximum tolerated dose (MTD) and/or phase II recommended dose (RP2D).
Maximum tolerated dose (MTD) | 21 days after first dose
  Phase Ib: Assess the incidence of dose-limiting toxicity (DLT), and determine the maximum tolerated dose (MTD) and/or phase II recommended dose (RP2D).
Phase II recommended dose (RP2D). | 21 days after first dose
  Phase Ib: Assess the incidence of dose-limiting toxicity (DLT), and determine the maximum tolerated dose (MTD) and/or phase II recommended dose (RP2D).
Objective Response Rate (ORR) | 24 weeks
  Phase II: Objective Response Rate (ORRW24) evaluated by the Independent Review Committee (IRC) based on RECIST 1.1.

SECONDARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 2 year
  Phase Ib: To determine the preliminary efficacy by evaluating the objective response rate (ORR) of F520 combined with lenvatinib in patients with advanced solid tumors (The last subject completed the 8th cycle of administration and completed the corresponding visits).
Maximum Plasma Concentration (Cmax） | 30 days (±7 days) after the last dose, early withdrawal or occurrence of SAE or grade ≥ 3 TRAE related to the study drug
  Phase Ib: To evaluate the pharmacokinetic characteristics of F520 and lenvatinib in patients with advanced solid tumors.
Objective response rate (ORR) | 24 weeks
  Phase II: The objective response rate evaluated by the investigator based on RECIST 1.1 (ORRW24).
PFS | through study completion, an average of 2 year
  Phase II: PFS evaluated by IRC and investigator based on RECIST.
PFS | through study completion, an average of 2 year
  Phase II: PFS evaluated by IRC and investigator based on iRECIST.
Adverse events | 30 days after the last dose
  Phase II: Evaluate the number and percent of patients with adverse events/adverse reactions and serious adverse events/severe adverse reactions in selected patients with advanced solid tumors treated with F520 combined with lenvatinib.
Adverse reactions | 30 days after the last dose
  Phase II: Evaluate the number and percent of patients with adverse events/adverse reactions and serious adverse events/severe adverse reactions in selected patients with advanced solid tumors treated with F520 combined with lenvatinib.
Serious adverse events | 30 days after the last dose
  Phase II: Evaluate the number and percent of patients with adverse events/adverse reactions and serious adverse events/severe adverse reactions in selected patients with advanced solid tumors treated with F520 combined with lenvatinib.
Severe adverse reactions | 30 days after the last dose
  Phase II: Evaluate the number and percent of patients with adverse events/adverse reactions and serious adverse events/severe adverse reactions in selected patients with advanced solid tumors treated with F520 combined with lenvatinib.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No